CLINICAL TRIAL: NCT03449394
Title: Effect of 4-session Metacognitive Training in Chinese Adult Outpatients With Schizophrenia Spectrum Disorders and Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Suzanne Ho-wai So, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCT2.0
Record Dates: First submitted 2018-01-23; First posted 2018-02-28 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Delusions; Depression
Keywords: Psychosis; Depression; Metacognition; Attribution; Emotions
MeSH Terms: conditions — Delusions; Depression; Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Delusions (Tx) (Active Comparator)
  Interventions: Other: Metacognitive Training
- Delusions (TAU) (No Intervention)
- Depression (Tx) (Active Comparator)
  Interventions: Other: Metacognitive Training
- Depression (TAU) (No Intervention)

INTERVENTIONS:
Other: Metacognitive Training — 4 sessions of Metacognitive Training using 4 treatment modules each targeting different cognitive biases
  Arms: Delusions (Tx); Depression (Tx)

SUMMARY:
Psychological studies have shown that individuals tend to attribute causes of positive and negative events differently. Specifically, individuals hold an internalising or externalising bias of attribution which, in the case of particular patient groups, was found to polarize to the extreme. Such extreme attributional styles have found to have a direct impact on emotions, leading to a waning course of psychiatric disorders. This project aims to further examine the theoretical links between attributions and emotions using a transdiagnostic approach, and the effect of a 4-session process-based intervention on attributional biases.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Clinical diagnosis of non-organic psychosis or major depressive disorder
* Presentation of delusions/a moderate level of depression

Exclusion Criteria:

* Clinical diagnosis of psychotic depression or depression with psychotic features
* Primary diagnosis of substance misuse or learning disability
* Participation of any cognitive/reasoning training program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Attributional style as measured by the Internal, Personal and Situational Attributions Questionnaire (IPSAQ) | 6 months
  IPSAQ consists of hypothetical scenarios. Participants are required to think of a single, most likely causal explanation to each of the hypothesized situations, and then to categorize this cause as being internal, external-personal or external-situational.
Psychotic symptomatology as measured by Positive and Negative Syndrome Scale (PANSS) | 6 months
  Positive and Negative Syndrome Scale (PANSS) is an interview-based assessment of the severity of symptoms associated with schizophrenia, including positive, negative, and general psychopathology.
Depressive symptomatology as measured by Beck Depression Inventory - II (BDI-II) and Calgary Depression Scale (CDS) | 6 months
  Beck Depression Inventory - II (BDI-II) is a 21-item self-report inventory that assesses symptoms of depression. Scores can range from 0 to 63, with higher scores reflecting greater symptom severity. Calgary Depression Scale (CDS) is a nine-item structured interview scale that assesses depressive symptoms in patients with schizophrenia.
Conviction of beliefs as measured by the Psychotic Symptom Rating Scale (PSYRATS) | 6 months
  The Psychotic Symptom Rating Scale (PSYRATS) is a 17-item semi-structured interview measuring the severity of multiple dimensions of auditory hallucinations and delusions, including conviction and duration.
Belief flexibility as measured by Maudsley Assessment of Delusions Schedule (MADS) and the BADE task | 6 months
  Maudsley Assessment of Delusions Schedule (MADS) is a standardised interview assessment that records whether participants could consider possibility of being mistaken (PM) about their delusional experience, any possible alternative explanations for the experience (EoE), and their reaction to hypothetical contradiction (RTHC). BADE task is an experimental design for measuring participants' bias against disconfirmatory evidence.
State-trait personality as measured by the State-Trait Personality Inventory (STPI) | 6 months
  State-Trait Personality Inventory (STPI) consists of 8 self-report scales, each containing 10 items covering state and trait anger, anxiety, curiosity and depression.

SECONDARY OUTCOMES:
Cognitive capacity as measured by the Chinese version of the Wechsler Adult Intelligence Scale - III (WAIS-III) | Baseline
  Three subtest short form - vocabulary, matrix reasoning and information - will be administered at baseline to assess the participants' cognitive capacity.
Severity of generalized anxiety disorder as measured by Generalised Anxiety Disorder 7 (GAD-7) | 6 months
  Generalised Anxiety Disorder 7 (GAD-7) is a self-reported questionnaire for screening and assessing severity of generalised anxiety disorder (GAD). This scale consists of seven items that measure severity of various signs of GAD according to reported response categories.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No